CLINICAL TRIAL: NCT06598891
Title: Effect of Combined PAS Balance Training on Individuals With PD
Brief Title: PAS Balance Training for Parkinson Disease (PD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PD_002
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: PD - Parkinson's Disease
Keywords: Gait Initiation; Paired associative stimulation (PAS); Balance training; Motor learning; Anticipatory postural adjustment (APA)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD APA training group (Experimental): Weight shift training and APA feedback.
  Interventions: Procedure: Weight shift training and APA feedback
- PD PAS group (Experimental): Using PAS to regulate brain plasticity
  Interventions: Procedure: Paired associative stimulation

INTERVENTIONS:
Procedure: Weight shift training and APA feedback — Use COP trajectory to train weight shift on force plate. To give APA visual feedback for subjects after weight shift training.
  Other Names: APA training
  Arms: PD APA training group
Procedure: Paired associative stimulation — Use TMS combine ES to stimulate TA nerve and M1 cortical
  Other Names: PAS training
  Arms: PD PAS group

SUMMARY:
Gait initiation (GI) difficulty is a common problem in individuals with Parkinson's disease (PD), often linked to impaired anticipatory postural adjustments (APA). Currently, there are no targeted rehabilitation programs designed specifically for GI-related APA in PD patients. Research has shown that while motor learning deficits are common in PD, explicit learning is better preserved than implicit learning. Therefore, a GI-related APA training system using an explicit learning model could be particularly effective for this population.

During motor learning, long-term potentiation (LTP) increases the excitability of the primary motor cortex. Paired associative stimulation (PAS) has been demonstrated to induce LTP-like changes in the motor cortex, making it a potential priming method to enhance motor learning. However, the priming effect of PAS targeted at leg muscles and the motor cortex on motor learning related to GI-APA has not been previously studied.

The objectives of this study are:

1. To investigate the effects of explicit and implicit training on GI-related APA.
2. To evaluate the priming effect of PAS on GI-related APA training and the associated plasticity changes in the motor cortex.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of Parkinson disease.

Exclusion Criteria:

* Musculoskeletal injuries on legs
* Osteoporosis.
* Any peripheral or central nervous system injury or disease patients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Balance Performance | Baseline, 4 weeks and 8 weeks
  Measured by the duration the stance or stand can be maintained. Unit：second(s)
COP Path Length in Balance Tasks | Baseline, 4 weeks and 8 weeks
  The total distance traveled by the COP over a specified period. Longer path lengths can indicate increased effort to maintain balance or greater instability.
COP Displacement in Balance Tasks | Baseline, 4 weeks and 8 weeks
  Measures of COP movement in the anterior-posterior (AP) and medial-lateral (ML) directions, offering insights into the directional tendencies of balance control. Unit：millimeter(mm)
Motor Evoked Potentials (MEPs) | Baseline, 4 weeks and 8 weeks
  MEPs are the electrical responses recorded from muscles following stimulation of the motor cortex. They reflect the efficiency of neural transmission from the cortex to the muscle. Unit：millivolts (mV)
Intracortical Facilitation (ICF) | Baseline, 4 weeks and 8 weeks
  ICF is measured by applying a pair of TMS pulses with a short interval (e.g., 8-15 ms) where the first (subthreshold) pulse is followed by a second (suprathreshold) pulse, leading to an increased amplitude of the MEP.
Intracortical Inhibition (ICI) | Baseline, 4 weeks and 8 weeks
  ICI is measured similarly to ICF but with a shorter inter-stimulus interval (e.g., 1-5 ms), resulting in a suppressed MEP amplitude. This suppression reflects inhibitory processes within the cortex.
Walking Speed | Baseline, 4 weeks and 8 weeks
  The time taken by participants to walk a standardized distance, typically expressed in centimeters per second (cm/s).
Step Length | Baseline, 4 weeks and 8 weeks
  The linear distance between the two ankles, typically expressed in centimeter(cm).
Step Time | Baseline, 4 weeks and 8 weeks
  The duration taken for one complete step, measuring from foot-off of one foot to the next foot-off of the same foot, usually expressed in seconds.

SECONDARY OUTCOMES:
COP Velocity in Balance Tasks | Baseline, 4 weeks and 8 weeks
  The speed at which the COP moves, calculated over the duration of the balance task. Higher velocities may reflect more dynamic balance adjustments or instability. Unit：millimeter per second(mm/s)
COP Area in Balance Tasks | Baseline, 4 weeks and 8 weeks
  The area covered by the COP trajectory during the balance task, providing an estimate of the sway envelope. A larger area might indicate poorer balance control. Unit：square millimeter(mm^2)
Double Support Time | Baseline, 4 weeks and 8 weeks
  The portion of the gait cycle where both feet are in contact with the ground, indicating the transition phase between steps, expressed as a percentage of the gait cycle or in seconds.
Single Support Time | Baseline, 4 weeks and 8 weeks
  The duration within the gait cycle when only one foot is in contact with the ground, typically measured in seconds or as a percentage of the total gait cycle.
Swing Time | Baseline, 4 weeks and 8 weeks
  The portion of the gait cycle where the foot is not in contact with the ground, moving forward to the next step. It is usually expressed as a percentage of the total gait cycle or in seconds.
Stance Time | Baseline, 4 weeks and 8 weeks
  The portion of the gait cycle when the foot is in contact with the ground, supporting body weight. It's typically expressed as a percentage of the total gait cycle or in seconds
Cadence | Baseline, 4 weeks and 8 weeks
  The number of steps an individual takes per minute, providing an overview of gait speed and rhythm, , expressed as steps per minute.

OTHER OUTCOMES:
Total UPDRS-III Score | Baseline
  The Unified Parkinson's Disease Rating Scale (UPDRS) Part III, also known as the UPDRS-III or the Motor Examination, is a critical component of the UPDRS used to assess the motor symptoms of Parkinson's disease (PD). To provide a comprehensive assessment of motor function in individuals with Parkinson's disease, covering aspects such as bradykinesia (slowness of movement), rigidity, tremors, and postural instability. The UPDRS-III consists of 14 items, each rated on a scale from 0 (normal) to 4 (severe), with a total possible score range from 0 to 108. Higher scores indicate greater motor impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan